CLINICAL TRIAL: NCT07084077
Title: Investigating the Effects of a Short Narratology Education Module on Empathy and Patient-centred Communication in Early-stage Medical Students: an Empirical Mixed-methods Pilot Study.
Brief Title: Investigating the Effects of a Short Narratology Education Module on Empathy and Patient-centred Communication in Early-stage Medical Students.
Status: Completed | Type: Observational
Sponsor: Connolly Hospital Blanchardstown (Other)
Responsible Party: Principal Investigator, Michael J Daly, MA MD PhD, Consultant Cardiologist, Senior Lecturer, Connolly Hospital Blanchardstown
Other Study IDs: REC202405007
Record Dates: First submitted 2025-07-17; First posted 2025-07-24 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Empathy; Patient-centredness; Narrative Medicine
Keywords: Empathy; Patient-centred communication; narrative medicine; medical education
MeSH Terms: conditions — Narrative Medicine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Narratology education module — At RCSI Dublin, mentioned by James Joyce in Dubliners, a one-week student-choice module Narrative Medicine: lessons from Irish writers and storytellers was offered to those in the second of our five-year undergraduate medical degree program, i.e., students were 18-months into the curriculum, had limited communication skills training, and no real-world clinical exposure. The module used close reading, group viewing, small-group workshops, and whole-group discussions to foster narrative competence. A medically-trained narratology-expert facilitated students' interrogation of classic and award-winning non-healthcare themed works by Irish writers and storytellers, i.e., directors and/or producers.

SUMMARY:
Effective communication is a fundamental skill in clinical medicine; however, traditional approaches often fail to equip learners with an ability to authentically and empathically engage with the complexities of real patients' experiences. Narratology education has been proposed as a pedagogical framework for augmenting empathy and patient-centred communication in medical students.

In April 2025, we undertook a mixed-methods pilot study to evaluate the impact of a one-week narratology education module on second-year undergraduate medical students at the Royal College of Surgeons in Ireland (RCSI), Dublin. The module involved close reading, group viewings, facilitated small-group workshops, and whole-group discussions in response to narrative works by Irish writers and storytellers, followed by written personal reflections. At the outset and conclusion of the module, each student undertook a clinical history with a simulated patient (SP) portraying early-stage dementia. SPs assessed each student's empathy and communication using the CARE Measure.

DETAILED DESCRIPTION:
Effective communication is a fundamental skill in clinical medicine; however, traditional approaches often fail to equip learners with an ability to authentically and empathically engage with the complexities of real patients' experiences. Narratology education has been proposed as a pedagogical framework for augmenting empathy and patient-centred communication in medical students.

In April 2025, we undertook a mixed-methods pilot study to evaluate the impact of a one-week narratology education module on second-year undergraduate medical students at the Royal College of Surgeons in Ireland (RCSI), Dublin. The module involved close reading, group viewings, facilitated small-group workshops, and whole-group discussions in response to narrative works by Irish writers and storytellers, followed by written personal reflections. At the outset and conclusion of the module, each student undertook a clinical history with a simulated patient (SP) portraying early-stage dementia. SPs assessed each student's empathy and communication using the CARE Measure.

Included students undertook two encounters with a simulated patient (SP): one immediately before and one immediately after the one-week narratology education module. In each encounter, students carried out a 7-minute history-taking exercise with an SP portraying cognitive decline/early-stage dementia. Immediately following each encounter, each SP completed the CARE Measure (11) - a validated tool to assess empathy and communication skills in healthcare workers. In the CARE Measure, ten items are rated on a five-point scale from 1 (poor) to 5 (excellent), with the total score being the sum of those ten items; in the event of missing or not applicable (N/A) ratings, the mean rating of available items was calculated and then multiplied by ten to estimate the total score. The CARE Measure items cover key aspects of empathy and clinical communication, including "Really listening," "Letting you tell your story," "Showing care and compassion," and "Being interested in you as a whole person." Ten SPs, with experience in medical education, were employed to perform a scripted-narrative of cognitive decline/early-stage dementia that had been iteratively developed by the investigating team and agreed by consensus prior to the start of the module. Each SP received the approved scripted-narrative one-week prior to the start of the module; in addition, they undertook a one-hour group pre-briefing session immediately prior to each simulation to ensure consistency of performance. Both pre-briefing sessions were facilitated by the investigating team including the narratology-expert.

At the end of the module, students submitted a reflective essay, i.e., 500-words using the Gibbs cycle as a framework, articulating how they had interrogated the narrative works of Irish writers and storytellers during the week and how narratology education had affected their appreciation for point-of-view and perspective in personal stories, their evolving narrative competence, and their empathy, communication, and performance in healthcare encounters.

Statistical analyses were undertaken using Stata/SE 17.0 (StataCorp [2021] Stata: Release 17. College Station, TX: StataCorp LLC.), GraphPad Prism version 10 (GraphPad Software, Boston, Massachusetts USA), and NVivo 15 (Lumivero [2023] NVivo (Version 15). Lumivero.).

Central tendencies for ordinal data are presented as median (interquartile range [IQR]). Pre- and post-intervention CARE Measure total scores and their individual item ratings were compared using the Wilcoxon matched-pairs signed-rank test, with a two-tailed P < 0.05 considered statistically significant.

Reflection essays were uploaded to NVivo 15 for thematic analysis.

ELIGIBILITY:
Inclusion Criteria:

Second-year medical students at RCSI Dublin Over 18 years of age Electing to take the student-choice module in Narrative Medicine

Exclusion Criteria:

English not as a first language

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Second-year medical students at RCSI Dublin
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2025-04-02 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-07-10 (Actual)

PRIMARY OUTCOMES:
Change in total Consultation and Relational Empathy (CARE) Measure score as assessed by Simulated Patients | 1 week
  In the CARE Measure, ten items are rated on a five-point scale from 1 (poor) to 5 (excellent), with the total score being the sum of those ten items (maximum score 50, minimum score zero); in the event of missing or not applicable (N/A) ratings, the mean rating of available items was calculated and then multiplied by ten to estimate the total score.
Change in individual Consultation and Relational Empathy (CARE) Measure score items' scores as assessed by Simulated Patients | 1 week
  In the CARE Measure, ten items are rated on a five-point scale from 1 (poor) to 5 (excellent), with the total score being the sum of those ten items (maximum score 50, minimum score zero); in the event of missing or not applicable (N/A) ratings, the mean rating of available items was calculated and then multiplied by ten to estimate the total score.

CONTACTS AND LOCATIONS:
Locations (1):
- RCSI School of Medicine, Dublin, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alhaidari B, Mulhall C, Condron C, Shpigelman J, Jain D, Daly MJ. Investigating the effects of a short narratology module on empathy and patient-centred communication in early-stage medical students: an empirical mixed-methods pilot study. BMC Med Educ. 2025 Dec 2;26(1):15. doi: 10.1186/s12909-025-08264-7. PMID 41331818